CLINICAL TRIAL: NCT05841199
Title: Coronary Epicardial and Microcirculatory Determinants of Ventricular Tachycardia Tolerability
Brief Title: Coronary Flow During Rapid Heart Rates
Acronym: VT flow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH7955
Record Dates: First submitted 2023-03-23; First posted 2023-05-03 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Ventricular Tachycardia; Coronary Artery Disease; Heart Failure; Coronary Microvascular Dysfunction; Coronary Microvascular Disease
Keywords: Ventricular Tachycardia; Coronary Artery Disease; Heart Failure; Coronary Microvascular Dysfunction; Coronary Microvascular Disease; Percutaneous Coronary Intervention; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular; Coronary Artery Disease; Heart Failure; Microvascular Angina | interventions — Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Controls: 10 patients with unobstructed coronary arteries, normal microvascular function and normal LV function.
  Interventions: Diagnostic Test: Pressure and flow measurement during simulated VT
- Coronary artery disease: 25 patients with severe, single-vessel coronary artery disease of the proximal LAD or proximal other dominant vessel awaiting PCI.
  Interventions: Diagnostic Test: Pressure and flow measurement during simulated VT
- Microvascular dysfunction: 15 patients with without severe disease in any coronary artery, impaired microvascular function and normal LV function.
  Interventions: Diagnostic Test: Pressure and flow measurement during simulated VT
- Heart failure: 20 patients with LV systolic dysfunction (LVEF<40%).
  Interventions: Diagnostic Test: Pressure and flow measurement during simulated VT

INTERVENTIONS:
Diagnostic Test: Pressure and flow measurement during simulated VT — Participants undergoing coronary angiography will have measurements of blood pressure, coronary pressure and coronary flow during simulated VT. VT will be simulated using pacing at a range of heart rates.

SUMMARY:
The goal of this observational study is to learn about the factors which determine how well ventricular tachycardia (VT) is tolerated. The main questions it aims to answer are:

1. What impact does coronary artery disease have on the ability for a patient to tolerate VT?
2. Does treatment of coronary artery disease with stents improve the tolerability of VT?

Participants who are undergoing a clinically indicated coronary angiogram or coronary angioplasty procedure will have measurements of blood pressure, coronary pressure and coronary flow made during pacing at a range of heart rates.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) is a common and life-threatening arrhythmia that occurs in people with heart problems. Some patients who develop this arrhythmia remain very stable with very little symptoms while others become unstable with low blood pressure or even sudden death. It is not known why some people tolerate the arrhythmia well and others do not.

If VT is not tolerated then current practice is to offer an implantable cardioverter defibrillator (ICD) which can deliver a shock to the heart if dangerous heart rhythms are detected. While shocks can be life-saving, they are also harmful, including causing psychological distress. ICDs also frequently deliver shocks when they are not needed.

If research could identify which factors predispose a person to be stable or unstable in VT, this would allow doctors to help them in a range of ways. One way would be to treat patients to improve the tolerance of VT, so avoiding the need for an ICD. Another would be to assess the the risk of instability and so allow a patient-centred decision on whether an ICD is needed.

In this study the investigators plan to recruit patients who are referred for a coronary angiogram. During the angiogram, the investigators will stimulate the heart at a range of fast heart rates and measure their blood pressure and flow in their coronary arteries. In patients who undergo stenting for a coronary stenosis, the investigators will also make these measurements after stenting so they can see if there is any difference. By recruiting a range of different cardiology patients, the investigators will be able to assess which factors contribute to stability during VT.

ELIGIBILITY:
Inclusion Criteria:

* Able to give valid consent
* Referred for coronary angiography or coronary angioplasty
* Suitable for percutaneous physiological interrogation and PCI when clinically indicated

Exclusion Criteria:

* Unable to give valid consent
* Pregnant or breastfeeding women
* Unstable coronary artery disease (acute coronary syndrome)
* Severe multivessel coronary artery disease suitable for coronary artery bypass grafting
* Severe heart valve disease
* Severe (NYHA IV) heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults referred for coronary angiography or coronary angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in coronary flow in participants with different levels of coronary microvascular function. | At baseline and during simulated VT
Change in coronary flow in participants immediately before and after PCI | At baseline and during simulated VT, immediately before PCI and after PCI
Change in blood pressure in participants with different levels of coronary microvascular function. | At baseline and during simulated VT
Change in blood pressure in participants before and after PCI | At baseline and during simulated VT, immediately before PCI and after PCI

SECONDARY OUTCOMES:
Change in coronary flow in participants with different levels of left ventricular function | At baseline and during simulated VT
Change in blood pressure in participants with different levels of left ventricular function | At baseline and during simulated VT

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Petraco, Principal Investigator — Senior Clinical Research Fellow
Locations (1):
- Imperial College NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided